CLINICAL TRIAL: NCT05558488
Title: Effect of a Meatless,Ketogenic Restrictive Diet on Body Composition, Concentration of Trimethylamine N-Oxide (TMAO),Ketone Bodies and Glucose in Blood and Urine, Somatic Disorders, Strength Capacity, Oxidative Stress, Immune Response
Brief Title: The Effect of a Meatless,Keto Restrictive Diet on Body Composition,Strength Capacity,Oxidative Stress,Immune Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Katarzyna Siedzik (Other)
Responsible Party: Sponsor-Investigator, Katarzyna Siedzik, Principal Investigator, Poznan University of Physical Education
Organization: Poznan University of Physical Education (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: KETOPROJEKT2019*2023
Record Dates: First submitted 2022-09-23; First posted 2022-09-28 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Body Weight; Oxidative Stress; Trimethylamine N-oxide; Immunologic Factors; Glucose Metabolism Disorders; Insulin Resistance; Insulin Sensitivity; Insulin Tolerance; Carbohydrate Metabolism Disorder; Lipid Metabolism Disorders; Body Fat Disorder; Ketosis; Ketoses, Metabolic; Somatic Disorders
Keywords: ketogenic diet; ketosis; oxidative stress; immune response; insulin resistance; body composition; strength capacity; omega 3 acids; meatless diet
MeSH Terms: conditions — Body Weight; Glucose Metabolism Disorders; Insulin Resistance; Lipid Metabolism Disorders; Ketosis

STUDY DESIGN:
Intervention Model Description: Each participant received a nutritional plan that was the same qualitatively but differed quantitatively. It was calculated for each individual based on the Mifflin-St Jeor Equation (Basal Metabolic Rate).
  After that, the levels of physical activity (PAL) were used to assess physical activity patterns and energy expenditure of individuals for placement into one of four PAL categories: sedentary, low active, active, or very active. That helped to calculate EER and made an individual reduction (minus 500 kcal / day). Before the start of the study, each participant obtained information about the basic principles of the ketogenic diet. Diet was designed to be isoproteic (1.8 g x Kg- 1 x body weight- 1 x day-1) with three meals a day. The distribution of macronutrients during the ketogenic diet (KD) was: protein 1.8 g x Kg-1 x body weight- 1 x day-1 (~ 25-30%), fats (~ 65-70%, with a strong emphasis on the content of omega 3 fatty acids) and carbohydrate (< 30 g x day- 1; < 10%).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Meatless restrictive ketogenic diet (Experimental): Diet was designed to be isoproteic (1.8 g x Kg- 1 x body weight- 1 x day-1) with three meals a day., restrictive (EER minus 500 kcal / day). The distribution of macronutrients during the very low carbohydrate ketogenic diet (KD) was: protein 1.8 g x Kg-1 x body weight- 1 x day-1 (~ 25-30%), fats (~ 65-70%, with a strong emphasis on the content of omega 3 fatty acids) and carbohydrate (< 30 g x day- 1; < 10%).
  Interventions: Other: Meatless, restrictive ketogenic diet

INTERVENTIONS:
Other: Meatless, restrictive ketogenic diet — Each participant received a nutritional plan that was the same qualitatively but differed quantitatively - a 500 kcal reduction based on Estimated Energy Requirement (EER) was assumed. Before the start of the study, each participant obtained information about the basic principles of the ketogenic diet. Diet was designed to be isoproteic (1.8gxKg-1xbody weight-1xday-1) with three meals a day. The distribution of macronutrients during the very low carbohydrate ketogenic diet (KD) was: protein 1.8 gxKg-1xbody weight-1xday-1(~25-30%), fats (~65-70%,with a strong emphasis on the content of omega 3 fatty acids) and carbohydrate (<30gxday-1;<10%).
  The food lists encouraged the consumption of fish,raw and cooked vegetables, eggs,fruits with the lowest glycemic index (blueberry, raspberry), plant oils and fats from avocado,olives.Drinks permitted were tea, coffee without sugar and the foods and drinks to be avoided were alcohol,meat (any kind of meat),bread,pasta,rice,milk,dairy and potatoes.

SUMMARY:
The subject of doctoral dissertation: Assessment of the effects of a meatless, ketogenic restrictive diet on body composition, strength capacity, oxidative stress and immune response

During planning of research and topic of the doctoral dissertation, it was considered how to modify a standard ketogenic diet rich in saturated fatty acids so that the use of this model of nutrition has the most anti-inflammatory effect. Therefore, it was decided to conduct a research to check whether a diet rich in omega-3 polyunsaturated fatty acids will show such an effect when following a high-fat diet.

Hypotheses:

1. The ketogenic diet reduces systemic inflammation. 2.The ketogenic diet reduces oxidative stress. 3. The ketogenic diet reduces body fat. 4. A ketogenic diet does not worsen strength performance.

DETAILED DESCRIPTION:
a) main research assumption

Reports in the international literature regarding the importance of the ketogenic diet are ambiguous. Some researchers believe that its use reduces body fat and improves insulin sensitivity or lipid profile, while others question this view and question it. Many authors emphasized the need for further research in this area, and this outline of the research project responds to this postulate.

In the presented experiment, the duration of a single experiment was 14 days, because the individual adaptation period of each participant should be taken into account - the so-called "keto-adaptation".

In order to assess the effectiveness of the nutritional intervention in this experiment, the following were performed: blood sampling for the determination of basic parameters (lipid profile, fasting glucose, fasting insulin, diabetic panel, hormones), determination of glucose and ketone bodies (β ketones) in the blood using a strip test - Optium Xido Neo glucometer, determination of the concentration of ketone bodies (acetoacetic acid) and glucose in the urine using Keto-Diastix - a strip test, examination by means of tests - force (maximum isokinetic force test with the use of Biodex apparatus), determination of inflammatory markers (TNF alpha, pro-inflammatory, anti-inflammatory and pro-or anti-inflammatory interleukins depending on the conditions), determination of oxidative stress markers - related to free radical damage to proteins (carbonyl groups, sulfhydryl groups (SH groups)), body composition measurement using the DEXA method (Dual Energy X-ray Absorptiometry). Choosing this method instead of the very common bioimpedance, due to the fact that using densitometry, it obtained very precise results of adipose tissue.

The above-described procedures were used to check the molecular basis of the phenomenon under study, to determine the parameters in which significant changes are visible and to determine the extent to which they translate into the function of the muscle and the subjective feelings of the subject.

Research methodology:

* body composition (DEXA)- Isometric muscle strength (Biodex)
* blood tests (lipid profile, glucose, insulin, ketone bodies)
* inflammatory markers - Luminex method with the use of BioRad BioPlex 200 reader Pro and anti-inflammatory cytokines (Bio-Plex Pro ™ Human Cytokine 8-plex Assay M50000007A, BIO-RAD, USA) (including IFN-y, IL-6, IL-8, IL-10, TNF-a, IL-2, IL-4)
* metabolic panel - Luminex method with the use of BioRad BioPlex 200 readerm (Bio-Plex Pro ™ Human Diabetes 10-Plex Assay # M171A7001M, BIO-RAD, USA) (including ghrelin, glucagon, insulin, leptin, resistin)
* markers of oxidative stress - Colorimetric method; Plate-based colorimetric measurement (360-385 nm) (concentration of protein carbonyl groups: Protein Carbonyl Colorimetric Assay Kit No. 100005020 (Cayman Chemical, Ann Arbor, MI, USA)
* markers of oxidative stress (concentration of protein thiol groups)
* TMAO (trimethylamine N-oxide)

ELIGIBILITY:
Inclusion Criteria:

* male or female
* healthy
* age 32 - 59
* non-smoker
* not abusing alcohol
* not subjected to physical exercise for at least 48 hours before the examination

Exclusion Criteria:

* cardiovascular,
* thyroid disease,
* gastrointestinal,
* respiratory
* or any other metabolic diseases adherence to special diets, use of nutritional supplements and use of medication to control blood lipids or glucose

Ages: 32 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Body composition | 2 weeks
  Whole body and regional body composition were measured in the morning after a 12 hours overnight fast by dual energy X-ray absorptiometry (DEXA) Body Composition: Body Fat Mass, Fat Free Mass, and Visceral Body Fat
  Body Fat Mass [Kg] max 40.143 Kg min 11.129 Kg (higher scores mean a worse outcome)
  Fat Free Mass [Kg] max 68.527 Kg min 37.72 Kg (higher scores mean a better outcome)
  Visceral Body Fat [g] max 2139 g min 90 g (higher scores mean a worse outcome)
Body weight | 2 weeks
  Body weight was measured with an accuracy of 0.1 Kg using an electronic scale (Tanita BC-601, Japan)
  Body weight (higher scores mean a worse outcome) [Kg] max 95.7 Kg min 60.9 Kg
TMAO | 2 weeks
  Trimethylamine N-Oxide (measured by Institute of Biochemistry and Biophysics Polish Academy of Sciences, Warsaw Poland)
  TMAO [ng/ml] (higher scores mean a worse outcome)
Lipids level (TC, HDL, LDL, TG) | 2 weeks
  Level of lipids - (TC- Total Cholesterol, LDL- low-density lipoprotein, HDL- high-density lipoprotein, TG - triacylglycerol)
  TC [mg/dl] (higher scores mean a worse outcome) LDL [mg/dl] (higher scores mean a worse outcome) TG [mg/dl] (higher scores mean a worse outcome) HDL [mg/dl] (higher scores mean a better outcome)
glucose level (blood, urine) | 2 weeks
  glucose level (blood, urine) - measured by Ketodiastix and Optimum Xido Neo
  higher scores mean a worse outcome
ketone bodies (blood, urine) | 2 weeks
  ketone bodies (blood, urine) - measured by Ketodiastix and Optimum Xido Neo
  higher scores mean a better outcome
inflammatory markers | 2 weeks
  inflammatory markers (including IFN-y, IL-6, IL-8, IL-10, TNF-a, IL-2, IL-4) - Luminex method with the use of BioRad BioPlex 200 reader Pro and anti-inflammatory cytokines (Bio-Plex Pro ™ Human Cytokine 8-plex Assay M50000007A, BIO-RAD, USA)
  depends - higher scores mean a better or worse outcome
markers of oxidative stress 1 | 2 weeks
  markers of oxidative stress - concentration of protein carbonyl groups - Colorimetric method; Plate-based colorimetric measurement (360-385 nm) (concentration of protein carbonyl groups: Protein Carbonyl Colorimetric Assay Kit No. 100005020 (Cayman Chemical, Ann Arbor, MI, USA)
  higher scores mean a worse outcome
markers of oxidative stress 2 | 2 weeks
  markers of oxidative stress - concentration of protein thiol group
  higher scores mean a worse outcome
metabolic panel - diabetes | 2 weeks
  metabolic panel - diabetes (including ghrelin, glucagon, insulin, leptin, resistin) - Luminex method with the use of BioRad BioPlex 200 readerm (Bio-Plex Pro ™ Human Diabetes 10-Plex Assay # M171A7001M, BIO-RAD, USA)
  depends - higher scores mean a better or worse outcome
somatic disorders | 2 weeks
  Somatic disorders measured by questionnaire based on Likert's scale
  Likert's scale:
  1. - Strongly disagree
  2. - Disagree
  3. - Neither agree nor disagree
  4. - Agree
  5. - Strongly agree
  It depends on question - higher scores mean a better or worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Katarzyna Siedzik, MSc, Principal Investigator — Poznan University of Physical Education, Poznan, Poland
Locations (1):
- Poznan University of Physical Education, Poznan, Greater Poland Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Phinney SD. Ketogenic diets and physical performance. Nutr Metab (Lond). 2004 Aug 17;1(1):2. doi: 10.1186/1743-7075-1-2. PMID 15507148
- [Background] Paoli A, Grimaldi K, Toniolo L, Canato M, Bianco A, Fratter A. Nutrition and acne: therapeutic potential of ketogenic diets. Skin Pharmacol Physiol. 2012;25(3):111-7. doi: 10.1159/000336404. Epub 2012 Feb 11. PMID 22327146
- [Background] Paoli A, Rubini A, Volek JS, Grimaldi KA. Beyond weight loss: a review of the therapeutic uses of very-low-carbohydrate (ketogenic) diets. Eur J Clin Nutr. 2013 Aug;67(8):789-96. doi: 10.1038/ejcn.2013.116. Epub 2013 Jun 26. PMID 23801097
- [Background] Paoli A, Bosco G, Camporesi EM, Mangar D. Ketosis, ketogenic diet and food intake control: a complex relationship. Front Psychol. 2015 Feb 2;6:27. doi: 10.3389/fpsyg.2015.00027. eCollection 2015. PMID 25698989
- [Background] Dashti HM, Mathew TC, Hussein T, Asfar SK, Behbahani A, Khoursheed MA, Al-Sayer HM, Bo-Abbas YY, Al-Zaid NS. Long-term effects of a ketogenic diet in obese patients. Exp Clin Cardiol. 2004 Fall;9(3):200-5. PMID 19641727
- [Background] Veech RL. The therapeutic implications of ketone bodies: the effects of ketone bodies in pathological conditions: ketosis, ketogenic diet, redox states, insulin resistance, and mitochondrial metabolism. Prostaglandins Leukot Essent Fatty Acids. 2004 Mar;70(3):309-19. doi: 10.1016/j.plefa.2003.09.007. PMID 14769489
- [Background] Balasse EO, Fery F. Ketone body production and disposal: effects of fasting, diabetes, and exercise. Diabetes Metab Rev. 1989 May;5(3):247-70. doi: 10.1002/dmr.5610050304. PMID 2656155